CLINICAL TRIAL: NCT03401112
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study of IMR-687 in Adult Patients With Sickle Cell Anaemia (Homozygous HbSS or Sickle-β0 Thalassemia)
Brief Title: A Study of IMR-687 in Adult Participants With Sickle Cell Anemia (Homozygous HbSS or Sickle-β0 Thalassemia)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Collaborators: Imara, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMR-SCD-102; 2017-000653-39 (EudraCT Number)
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IMR-687 50 mg/100 mg (Experimental): A starting dose of IMR-687 50 mg with dose escalation after 4 or 12 weeks, up to 100 mg was administered to participants. Duration of administration was 16 (Week 17) or 24 weeks (Week 25).
  Interventions: Drug: IMR-687
- IMR-687 100 mg/200 mg (Experimental): A starting dose of IMR-687 100 mg with dose escalation after 4 or 12 weeks, up to 200 mg was administered to participants. Duration of administration was 24 weeks (Week 25).
  Interventions: Drug: IMR-687
- Placebo (Placebo Comparator): Matching placebo was administered for 16 (Week 17) or 24 weeks (Week 25).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMR-687 — Oral administration of IMR-687 once daily with or without HU.
  Arms: IMR-687 100 mg/200 mg; IMR-687 50 mg/100 mg
Drug: Placebo — Oral administration of placebo once daily with or without HU.
  Arms: Placebo

SUMMARY:
Study of IMR-687 in adult participants with sickle cell anemia (SCA) (homozygous HbSS or sickle-β0 thalassemia).

DETAILED DESCRIPTION:
This is a proof-of-concept study in adult SCA participants, ages 18 to 55 years old, to examine the safety, tolerability, and pharmacokinetic (PK), as well as the potential pharmacodynamic (PD) effects and clinical efficacy, of IMR-687 across a range of doses.

IMR-687 was administered in 2 populations of participants with SCA: those who were not receiving hydroxyurea (HU) and those who were receiving a stable dose of HU according to standard of care.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants with confirmed SCA
* Age 18 to 55 years, inclusive
* For participants on HU, must have been on a stable dose for at least 60 days prior to screening

Key Exclusion Criteria:

* Total hemoglobin >12.5 or <6 grams/deciliter
* Red blood cell transfusion within 60 days of baseline
* >7 hospitalizations for vaso-occlusive crises (VOCs) within the last year
* Estimated glomerular filtration rate <50 milliliter/minute
* Aspartate aminotransferase/alanine aminotransferase >3x the upper limit of normal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regulatory Operations, Study Director — Cardurion Pharmaceuticals
Locations (13):
- United States (7):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - University of Illinois, Chicago, Illinois
  - Loretto Hospital, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott & White Health, Temple, Texas
- United Kingdom (6):
  - Sandwell & West Birmingham Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Royal London Hospital, London
  - University College London Hospital, London
  - Guy's Hospital, London
  - Oxford Cancer & Haematology Centre, The Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled at 13 sites in 2 countries (United Kingdom and United States).
Groups:
- IMR-687 50 mg/100 mg (Without HU): A starting dose of IMR-687 50 milligrams (mg) with dose escalation after 4 or 12 weeks, up to 100 mg was administered to participants who were not receiving daily hydroxyurea (HU).
- IMR-687 100 mg/200 mg (Without HU): A starting dose of IMR-687 100 mg with dose escalation after 4 or 12 weeks, up to 200 mg was administered to participants who were not receiving daily HU.
- Placebo (Without HU): Matching placebo was administered to participants who were not receiving daily HU.
- IMR-687 50 mg/100 mg (With HU): A starting dose of IMR-687 50 mg with dose escalation after 4 or 12 weeks, up to 100 mg was administered to participants who were receiving daily HU. HU doses ranged from 500 to 2000 mg.
- Placebo (With HU): Matching placebo was administered to participants who were receiving daily HU. HU doses ranged from 500 to 2000 mg.
Period: Overall Study
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU) | Placebo (Without HU) | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU)
Started | 15 | 26 | 22 | 27 | 10
Received at Least 1 Dose of Study Drug | 12 | 26 | 20 | 25 | 10
Completed | 10 | 19 | 11 | 21 | 10
Not Completed | 5 | 7 | 11 | 6 | 0
Not completed — Adverse Event | 1 | 2 | 3 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Noncompliance | 1 | 2 | 3 | 0 | 0
Not completed — Did not Meet Inclusion Criteria | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0
Not completed — Study was Terminated by Sponsor | 0 | 0 | 0 | 1 | 0
Not completed — Day 1 Assessment not Done | 1 | 0 | 0 | 0 | 0
Not completed — Not Dosed | 0 | 0 | 1 | 0 | 0
Not completed — Missed Clinical Visit | 0 | 0 | 1 | 0 | 0
Not completed — Missed Doses | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who had received any amount of study drug.
Groups:
- IMR-687 50 mg/100 mg (Without HU): A starting dose of IMR-687 50 mg with dose escalation after 4 or 12 weeks, up to 100 mg was administered to participants who were not receiving daily HU.
- Total: Total of all reporting groups
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU) | Placebo (Without HU) | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU) | Total
Number analyzed (Participants) | 12 | 26 | 20 | 25 | 10 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (8.7) | 32.0 (9.3) | 35.2 (8.4) | 32.4 (9.1) | 28.8 (7.1) | 32.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 12 | 15 | 9 | 61
  Male | 4 | 9 | 8 | 10 | 1 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 11 | 23 | 19 | 24 | 9 | 86
  Not Reported | 1 | 1 | 0 | 1 | 0 | 3
  Unknown Ethnicity | 0 | 2 | 1 | 0 | 1 | 4
  Black or African American | 12 | 25 | 19 | 24 | 9 | 89
  Other | 0 | 1 | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Treatment-emergent Adverse Events (TEAEs) And Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An SAE was defined as any AE that resulted in 1 or more of the following outcomes: death, required or prolonged hospitalization, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, or other medically important event. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through up to Week 24
Population: All participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- All IMR-687: All participants who received IMR-687.
- All Placebo: All participants who received placebo.
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU) | Placebo (Without HU) | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU) | All IMR-687 | All Placebo
Number analyzed (Participants) | 12 | 26 | 20 | 25 | 10 | 63 | 30
Participants
  TEAEs | 12 | 24 | 18 | 23 | 10 | 59 | 28
  SAEs | 4 | 7 | 8 | 5 | 3 | 16 | 11

2. Secondary Outcome: Pharmacokinetic (PK) Of Participants Who Did Not Concomitantly Receive HU: Maximum Plasma Concentration (Cmax) Of IMR-687
Description: For PK assessments of participants who did not concomitantly receive HU, serial blood samples for IMR-687 plasma concentrations were drawn predose at 0.5, 1, 1.5, 2, 4, 6, and 8 hours after administration of study drug; and at 24 hours after administration of study drug. Day 1 (single-dose) and steady-state (Week 25) assessments are presented.
Time Frame: Day 1 and Week 25
Population: PK Analysis population consisted of all participants with sufficient sampling for PK parameter evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU)
Number analyzed (Participants) | 12 | 13
ng/mL
  Day 1: Single Dose | 512 (30.1) | 1130 (33.5)
  Week 25: Steady State: number analyzed (Participants) | 8 | 8
  Week 25: Steady State | 1290 (36.4) | 2180 (24.1)

3. Secondary Outcome: PK Of Participants Who Did Not Concomitantly Receive HU: Area Under The Concentration-time Curve (AUC) From Time 0 To 24 Hours Postdose (AUC0-24h) Of IMR-687
Description: as for outcome 2
Time Frame: Day 1 and Week 25
Population: PK Analysis population consisted of all participants with sufficient sampling for PK parameter evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU)
Number analyzed (Participants) | 11 | 10
h*ng/mL
  Day 1: Single Dose | 2850 (12.5) | 6590 (17.7)
  Week 25: Steady State: number analyzed (Participants) | 7 | 6
  Week 25: Steady State | 8420 (24.1) | 15000 (22.3)

4. Secondary Outcome: PK Of Participants Who Concomitantly Received HU: Cmax Of IMR-687
Description: For PK assessments of participants who concomitantly received HU, serial blood samples for IMR-687 PK were drawn predose at 0.5, 1, 1.5, 2, 4, 6, and 8 hours after administration of study drug; and at 24 hours after administration of study drug. Day 1 (single-dose) and steady-state (Week 17) assessments are presented.
Time Frame: Day 1 and Week 17
Population: PK Analysis population consisted of all participants with sufficient sampling for PK parameter evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IMR-687 50 mg/100 mg (With HU)
Number analyzed (Participants) | 13
ng/mL
  Day 1: Single Dose | 657 (24.7)
  Week 17: Steady State: number analyzed (Participants) | 8
  Week 17: Steady State | 1370 (18.6)

5. Secondary Outcome: PK Of Participants Who Concomitantly Received HU: AUC0-24h Of IMR-687
Description: For PK assessments of participants who concomitantly received HU, serial blood samples for IMR-687 plasma concentrations were drawn predose at 0.5, 1, 1.5, 2, 4, 6, and 8 hours after administration of study drug; and at 24 hours after administration of study drug. Day 1 (single-dose) and steady-state (Week 17) assessments are presented.
Time Frame: Day 1 and Week 17
Population: PK Analysis population consisted of all participants with sufficient sampling for PK parameter evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | IMR-687 50 mg/100 mg (With HU)
Number analyzed (Participants) | 12
h*ng/mL
  Day 1: Single Dose | 3090 (34.0)
  Week 17: Steady State: number analyzed (Participants) | 8
  Week 17: Steady State | 7300 (16.1)

6. Secondary Outcome: PK Of Participants Who Concomitantly Received HU: Cmax Of HU
Description: For PK assessments of participants who concomitantly received HU, serial blood samples for HU PK were drawn predose and at 0.5, 1, 1.5, 3, 6, 8, and 10 hours after self-administration of the prescribed dose of HU. HU in the presence (end of treatment [EOT]: Week 17) or absence of IMR-687 (Baselines 1 and 2) are presented. HU concentration data were not sorted with respect to HU dose.
Time Frame: Baseline (1 and 2) and Week 17
Population: PK Analysis population consisted of all participants with sufficient sampling for PK parameter evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- IMR-687 50 mg/100 mg (With HU): A starting dose of IMR-687 50 mg with dose escalation after 4 or 12 weeks, up to 100 mg was administered to participants who were also receiving daily HU. HU doses ranged from 500 to 2000 mg.
- Placebo (With HU): Participants who were receiving daily HU were administered placebo. HU doses ranged from 500 to 2000 mg.
Arm/Group | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU)
Number analyzed (Participants) | 14 | 6
μg/mL
  Baseline 1 | 25.3 (36.7) | 20.6 (87.8)
  Baseline 2 | 24.8 (38.1) | 25.4 (98.6)
  Week 17: number analyzed (Participants) | 10 | 5
  Week 17 | 24.5 (55.2) | 20.5 (127)

7. Secondary Outcome: PK Of Participants Who Concomitantly Received HU: AUC0-24h Of HU
Description: For PK assessments of participants who concomitantly received HU, serial blood samples for HU PK were drawn predose and at 0.5, 1, 1.5, 3, 6, 8, and 10 hours after self-administration of the prescribed dose of HU. HU in the presence (EOT: Week 17) or absence of IMR-687 (Baselines 1 and 2) are presented. HU concentration data were not sorted with respect to HU dose.
Time Frame: Baseline (1 and 2) and Week 17
Population: PK Analysis population consisted of all participants with sufficient sampling for PK parameter evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μg/mL
Arm/Group | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU)
Number analyzed (Participants) | 12 | 5
h*μg/mL
  Baseline 1: number analyzed (Participants) | 11 | 4
  Baseline 1 | 99.2 (32.4) | 113 (87.7)
  Baseline 2 | 103 (30.7) | 129 (71.7)
  Week 17: number analyzed (Participants) | 8 | 4
  Week 17 | 122 (23.0) | 91.4 (127)

8. Other Pre Specified Outcome: Change From Baseline In F-Cells
Description: Absolute least squares (LS) mean change from baseline at EOT is presented. Change from baseline in pharmacodynamic (PD) biomarkers was analyzed using mixed models for repeated measures with covariate of treatment, visit, treatment-by-visit interaction, and baseline value.
Time Frame: Baseline, EOT (Week 25 for participants without HU and Weeks 17 or 25 for participants with HU)
Population: All participants who had samples for PD analysis sufficient to obtain at least 1 valid PD observation, without protocol deviations or events that would be expected to affect the PD analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of F-cells
Groups:
- Pooled IMR-687 (Without HU): All participants administered IMR-687 who were not receiving daily HU.
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU) | Pooled IMR-687 (Without HU) | Placebo (Without HU) | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU)
Number analyzed (Participants) | 7 | 13 | 20 | 7 | 5 | 1
percentage of F-cells | 3.97 (4.07) | 5.66 (2.87) | 4.81 (2.48) | -6.00 (3.77) | -2.49 (6.00) | 7.38 (15.54)

9. Post Hoc Outcome: Number Of Participants With Vaso-occlusive Crisis (VOCs)
Description: VOCs include the events of acute painful crisis and acute chest symptoms (includes fever, cough, sputum production, shortness of breath, tachypnea, hypoxia, and chest pain).
Time Frame: Day 1 (after dosing) through up to Week 24
Population: All participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU) | Placebo (Without HU) | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU) | All IMR-687 | All Placebo
Number analyzed (Participants) | 12 | 26 | 20 | 25 | 10 | 63 | 30
Participants | 6 | 14 | 14 | 10 | 7 | 30 | 21

10. Post Hoc Outcome: Time To First VOC Event
Description: VOCs include the events of acute painful crisis and acute chest symptoms (includes fever, cough, sputum production, shortness of breath, tachypnea, hypoxia, and chest pain). Time to first VOC event was assessed by Kaplan Meier analysis. For this analysis, HU and without HU population groups were pooled for IMR-687 and placebo. In addition, pooled IMR-687 (all doses) are presented.
Time Frame: Day 1 (after dosing) through up to Week 24
Population: Pooled data from the IMR-687 dose groups (IMR-687 50mg/100 mg [Without HU]+ IMR-687 100mg/200 mg [Without HU] + IMR-687 50mg/100 mg [With HU]) and pooled data from the placebo arms (With and without HU) were used to provide a larger sample size for the analysis of time to 1st event.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- IMR-687 50 mg/100 mg: All participants who had a starting dose of IMR-687 50 mg (with HU and without HU) with dose escalation up to 100 mg was administered.
- IMR-687 100 mg/200 mg: All participants who had a starting dose of IMR-687 100 mg with dose escalation up to 200 mg was administered.
Arm/Group | IMR-687 50 mg/100 mg | IMR-687 100 mg/200 mg | All IMR-687 | All Placebo
Number analyzed (Participants) | 37 | 26 | 63 | 30
days | NA [60.00 to NA] — The median and upper confidence limit were non-estimable due to insufficient number of participants with an event to estimate variability and build a confidence interval. | 139.00 [35.00 to NA] — The upper confidence limit was non-estimable due to insufficient number of participants with an event to estimate variability and build a confidence interval. | 169.00 [80.00 to NA] — The upper confidence limit was non-estimable due to insufficient number of participants with an event to estimate variability and build a confidence interval. | 87.00 [26.00 to 167.00]
Statistical Analysis 1: Comparison: IMR-687 50 mg/100 mg vs IMR-687 100 mg/200 mg vs All Placebo; Test type: Superiority; p = 0.0686, Log Rank
Statistical Analysis 2: Comparison: All IMR-687 vs All Placebo; Test type: Superiority; p = 0.0294, Log Rank

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through up to Week 24
Description: Adverse event data are presented for each of the following IMR-687 groups which included a brief dose escalation: IMR-687 50mg/100 mg [Without HU], IMR-687 100mg/200 mg [Without HU], IMR-687 50mg/100 mg [With HU] and for each placebo arm. Data are not available by dose escalation within arms.
Arm/Group | IMR-687 50 mg/100 mg (Without HU) | IMR-687 100 mg/200 mg (Without HU) | Placebo (Without HU) | IMR-687 50 mg/100 mg (With HU) | Placebo (With HU) | All IMR-687 | All Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/26 | 0/20 | 0/25 | 0/10 | 0/63 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/12 | 7/26 | 8/20 | 5/25 | 3/10 | 16/63 | 11/30
Other Adverse Events (participants affected / at risk) | 12/12 | 22/26 | 16/20 | 23/25 | 10/10 | 57/63 | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IMR-687 50 mg/100 mg (Without HU) (N=12) | IMR-687 100 mg/200 mg (Without HU) (N=26) | Placebo (Without HU) (N=20) | IMR-687 50 mg/100 mg (With HU) (N=25) | Placebo (With HU) (N=10) | All IMR-687 (N=63) | All Placebo (N=30)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 3 (4) | 7 (8) | 7 (11) | 3 (3) | 3 (3) | 13 (15) | 10 (14)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/8 (1) | 0/17 (0) | 0/12 (0) | 0/15 (0) | 0/9 (0) | 1/40 (1) | 0/21 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/8 (0) | 0/17 (0) | 0/12 (0) | 1/15 (1) | 0/9 (0) | 1/40 (1) | 0/21 (0)
Rash generalise (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMR-687 50 mg/100 mg (Without HU) (N=12) | IMR-687 100 mg/200 mg (Without HU) (N=26) | Placebo (Without HU) (N=20) | IMR-687 50 mg/100 mg (With HU) (N=25) | Placebo (With HU) (N=10) | All IMR-687 (N=63) | All Placebo (N=30)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 5 (15) | 9 (15) | 9 (14) | 10 (14) | 6 (23) | 24 (44) | 15 (37)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 8 (14) | 0 (0) | 4 (4) | 5 (5) | 14 (21) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (3) | 0 (0) | 5 (7) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (4) | 5 (5) | 1 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (6) | 2 (2) | 7 (9) | 4 (4)
Influenza like illness (General disorders) | 2 (2) | 2 (3) | 2 (2) | 2 (5) | 0 (0) | 6 (10) | 2 (2)
Pain (General disorders) | 2 (2) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 4 (5) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ocular icterus (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 7 (7) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (2) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (1) | 2 (2) | 2 (3) | 2 (2) | 6 (9) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 2 (2) | 1 (1) | 2 (2) | 7 (8) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 6 (7) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 5 (6) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 8 (11) | 4 (6) | 12 (18) | 4 (6) | 22 (31) | 8 (12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03401112/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03401112/SAP_001.pdf